CLINICAL TRIAL: NCT03543462
Title: Diaphragmatic Resection And Gynecological Ovarian Neoplasm
Acronym: DRAGON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Head of Department of Women's and Children's Health, Policlinico Agostino Gemelli Foundation University Hospital, Rome, Italy, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D.R.A.G.O.N. ID. 1963
Record Dates: First submitted 2018-03-21; First posted 2018-06-01 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Diaphragm; Chest Drain; Diaphragmatic Resection; Pleural Effusion
MeSH Terms: conditions — Ovarian Neoplasms; Pleural Effusion

STUDY DESIGN:
Intervention Model Description: Patients affected by advanced stage ovarian cancer with diaphragmatic involvement. When diaphragmatic resection is performed the patients are randomized to proceed with chest drain positioning or not
Who Masked: Investigator
Masking Description: The investigator check the random list only when the patients is enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Chest tube positioning YES (Sham Comparator): Patients enrolled for chest tube positioning
  Interventions: Device: thoracic Drain Tube 24 Fr.
- Arm B: Chest tube positioning NO (No Intervention): Patients enrolled for diaphragm closure without chest tube positioning

INTERVENTIONS:
Device: thoracic Drain Tube 24 Fr. — Positioning of Thoracic Drain after diaphragmatic resection and consequently diaphragmatic repair
  Arms: Arm A: Chest tube positioning YES

SUMMARY:
Prospective randomized phase IV study aimed to value the impact of diaphragmatic surgery and the useful of intra-operatory thoracic drain in advanced ovarian cancer.

Considering the fact that the diaphragmatic surgery could contribute with the incidence of post-operatory morbidity. The study is aimed to value the role of thoracic drain in post-operative outcomes as hospital stay, time to chemotherapy, drugs use and eventual interventions.

DETAILED DESCRIPTION:
Ovarian cancer represents the leading cause of death from gynecologic malignancies. The majority of patients present with advanced-stage disease (III/IV) often involving the upper abdomen. Spread by either direct extension or via peritoneal implantation can result in metastases to the diaphragm, as seen in up to 40% of patients with advanced disease.

Standard treatment of advanced-stage disease includes primary cytoreductive surgery followed by combination platinum-taxane chemotherapy. Optimal cytoreduction to ≤1 cm disease has repeatedly been shown to be associated with improved survival.

Diaphragm involvement was considered one of the most frequent obstacles to achieving optimal cytoreduction. The right diaphragm is more frequently and extensively involved than the left diaphragm; however, bilateral involvement is not uncommon. Various studies have advocated and reported the feasibility of diaphragmatic surgery in achieving optimal cytoreduction.

Sometimes, depending on extent of the disease, the diaphragm involvement could be massive and often the resection of the muscle with access to pleural cavity is necessary. Allegedly, entering the pleural cavity increases the morbidity of the procedure.

Extensive upper abdominal surgery involving diaphragmatic peritonectomy/resection and liver mobilization may both contribute to the development of symptomatic pleural effusions.

The aim of the study is to value the impact of diaphragmatic surgery in post-operative complications using a specific score (DRS). The other aim is to asses a correct management of intra-operatory thoracic drain position after diaphragmatic surgery. All parameter that could influence the post-operative outcomes as (EBL,BMI, OT, SCS) are recorded.

The study was approved by Ethical Committee of Fondazione Policlinico Gemelli Hospital (prot n. 9078/18).

The study is a superiority randomized clinical trial to investigate the role of intra-operative chest tube in the large (> 5 cm) diaphragmatic peritonectomy/resection in the ovarian cancer debulking. Calculation of sample size for the analysis of the primary end-point (major pleural effusion) was based on literature results reporting a rate of moderate/severe early peri-operative pleural effusion between 54% and 23% when a large (> 5 cm) diaphragmatic resection is performed. A sample size of 88 patients was required in order to provide 80% power of detecting a reduction of 60% of moderate/severe pleural effusion in PDS with large diaphragmatic resection when intra-operative chest tube was inserted (overall rate 22%) (two-tailed α =0.05, drop-out 5%).

Sample size is composed by 44 Patients affected by advanced stage ovarian cancer, meeting inclusion criteria, undergo diaphragmatic surgery followed by intra-operatory thoracic drain position and 44 patients with same characteristics undergo to diaphragmatic surgery without intra-operatory thoracic drain position. Both groups are compared in terms of incidence of post-operative complications (especially pleural effusion, pneumothorax, respiratory disease). Secondary endpoints are the evaluation of surgical outcomes and clinical outcomes in terms hospital stay, procedures and radiologic examinations required. All patients are adequately informed and inserted in the study only after having read and signed an informed consent. Diagnostic, clinical and surgical data of each patient are prospectively recorded.

Surgical procedures consist of surgical standard cytoreduction, performed for all cases of advanced stage ovarian cancer disease. The procedures performed depending on disease spread.

The diaphragmatic procedures, depending on the disease infiltration can consists of superficial peritonectomy, deep peritonectomy (until muscular layer) or diaphragmatic resection. Considering the randomization, if required, a thoracic drain tube 24 Fr. is positioned. A post-operative chest X-Ray is performed on all cases.

At the end of the procedure, a schedule is compiled with intraoperative data.

Post-operative examinations are follows:

* Chest X-Ray (2 h post-op)
* Chest X-Ray (day 1)
* Chest X-Ray (if required, depending of clinical indications)
* Thoracic US scan evaluation before discharge
* Thoracic US scan evaluation 10 days after discharge
* Radiological examinations (if required, depending of clinical indications)

All clinical and histologic data will be recorded prospectively using an electronic database.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 < 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* No actual pregnancies or pelvic inflammatory disease (P.I.D.)
* BMI < 40
* Macroscopic diaphragmatic disease infiltration (mono lateral)
* Grade IIIA-IV diaphragmatic resection score
* Advanced stage ovarian cancer (stage III-IV)
* Primary diagnosis, interval debulking surgery, recurrent disease
* All histotype included

Exclusion Criteria:

* Actual pregnancies or P.I.D
* BMI > 40
* Pulmonary or thoracic preoperatory disease
* Preoperative pleural effusion
* Residual thoracic disease after surgery
* Residual diaphragmatic disease after surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Measurement of incidence of pleural effusion after diaphragmatic resection and useful of chest drain to prevent pleural effusion and consequent respiratory symptoms as dyspnea. | 30 days
  The diaphragmatic surgery is often related to post-operative complication. The most common complication is pleural effusion. This condition contribute to decrease the clinical outcomes causing increase of hospitalization and necessity medical or surgical treatment.
  The main outcome is to asses a correct management of intra-operatory thoracic drain position after diaphragmatic surgery.
  The outcomes measured are:
  - Incidence of post-operatory pleural effusion detected by chest RX measuring pleural fluid collection (cm)

OTHER OUTCOMES:
Time to start chemotherapy | 40 Days
  The time to start chemotherapy is fundamental from oncological point of view. The ideal time to start chemotherapy treatment should exceed 40 days after surgery.
  The data measured are
  - time between surgery and first chemotherapy cycle
Estimated blood loss | 1 Day
  The intra operative blood loss is often related to the complexity of procedure and consequently to post-operative complications
  The data measured are:
  - EBL (ml)
Operative time | 1 Day
  The Operative time is often related to the complexity of procedure and consequently to post-operative complications
  The data measured are:
  - Operative time (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cianci, M.D., Principal Investigator — Fondazione Policlinico Agostino Gemelli
Locations (1):
- Fondazione Policlinico Agostino Gemelli, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Eisenkop SM, Spirtos NM. What are the current surgical objectives, strategies, and technical capabilities of gynecologic oncologists treating advanced epithelial ovarian cancer? Gynecol Oncol. 2001 Sep;82(3):489-97. doi: 10.1006/gyno.2001.6312. PMID 11520145
- [Background] Bristow RE, Tomacruz RS, Armstrong DK, Trimble EL, Montz FJ. Survival effect of maximal cytoreductive surgery for advanced ovarian carcinoma during the platinum era: a meta-analysis. J Clin Oncol. 2002 Mar 1;20(5):1248-59. doi: 10.1200/JCO.2002.20.5.1248. PMID 11870167
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Carlson JW, Ozols RF, Rose PG, Markman M, Armstrong DK, Muggia F, McGuire WP; Gynecologic Oncology Group Study. Prognostic factors for stage III epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Aug 20;25(24):3621-7. doi: 10.1200/JCO.2006.10.2517. PMID 17704411
- [Background] Aletti GD, Dowdy SC, Podratz KC, Cliby WA. Surgical treatment of diaphragm disease correlates with improved survival in optimally debulked advanced stage ovarian cancer. Gynecol Oncol. 2006 Feb;100(2):283-7. doi: 10.1016/j.ygyno.2005.08.027. Epub 2005 Sep 22. PMID 16182350
- [Background] Tsolakidis D, Amant F, Van Gorp T, Leunen K, Neven P, Vergote I. The role of diaphragmatic surgery during interval debulking after neoadjuvant chemotherapy: an analysis of 74 patients with advanced epithelial ovarian cancer. Int J Gynecol Cancer. 2010 May;20(4):542-51. doi: 10.1111/IGC.0b013e3181d4de23. PMID 20686373
- [Background] Zapardiel I, Peiretti M, Zanagnolo V, Biffi R, Bocciolone L, Landoni F, Aletti G, Colombo N, Maggioni A. Diaphragmatic surgery during primary cytoreduction for advanced ovarian cancer: peritoneal stripping versus diaphragmatic resection. Int J Gynecol Cancer. 2011 Dec;21(9):1698-703. doi: 10.1097/IGC.0b013e31822f65c3. PMID 22080893
- [Background] Fanfani F, Fagotti A, Gallotta V, Ercoli A, Pacelli F, Costantini B, Vizzielli G, Margariti PA, Garganese G, Scambia G. Upper abdominal surgery in advanced and recurrent ovarian cancer: role of diaphragmatic surgery. Gynecol Oncol. 2010 Mar;116(3):497-501. doi: 10.1016/j.ygyno.2009.11.023. Epub 2009 Dec 11. PMID 20004958
- [Background] Chereau E, Ballester M, Selle F, Cortez A, Pomel C, Darai E, Rouzier R. Pulmonary morbidity of diaphragmatic surgery for stage III/IV ovarian cancer. BJOG. 2009 Jul;116(8):1062-8. doi: 10.1111/j.1471-0528.2009.02214.x. Epub 2009 May 14. PMID 19459863
- [Background] Devolder K, Amant F, Neven P, van Gorp T, Leunen K, Vergote I. Role of diaphragmatic surgery in 69 patients with ovarian carcinoma. Int J Gynecol Cancer. 2008 Mar-Apr;18(2):363-8. doi: 10.1111/j.1525-1438.2007.01006.x. PMID 18334014
- [Background] Eisenhauer EL, D'Angelica MI, Abu-Rustum NR, Sonoda Y, Jarnagin WR, Barakat RR, Chi DS. Incidence and management of pleural effusions after diaphragm peritonectomy or resection for advanced mullerian cancer. Gynecol Oncol. 2006 Dec;103(3):871-7. doi: 10.1016/j.ygyno.2006.05.023. Epub 2006 Jul 3. PMID 16815536
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Cliby W, Dowdy S, Feitoza SS, Gostout BS, Podratz KC. Diaphragm resection for ovarian cancer: technique and short-term complications. Gynecol Oncol. 2004 Sep;94(3):655-60. doi: 10.1016/j.ygyno.2004.04.032. PMID 15350355